CLINICAL TRIAL: NCT05977972
Title: Pattern of Metabolic Causes of Neonatal Hypoglycemia at Assiut University Children's Hospital
Brief Title: Pattern of Metabolic Causes of Neonatal Hypoglycemia
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Amany Mohammed Bakry Hassan, Principal Investigator, Assiut University
Other Study IDs: Neonatal hypoglycemia
Record Dates: First submitted 2023-07-24; First posted 2023-08-07 (Actual); Last update posted 2023-08-07 (Actual); Status verified 2023-07

CONDITIONS: Neonatal Hypoglycemia; Metabolic Disease
MeSH Terms: conditions — Metabolic Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective

SUMMARY:
Inborn errors of metabolism (IEM) are disorders in which there is a block at some point in the normal metabolic pathway caused by a genetic defect of a specific enzyme. The number of diseases in humans known to be attributable to inherited point defects in metabolism now exceeds 500.While the diseases individually are rare, they collectively account for a significant proportion of neonatal and childhood morbidity and mortality. Diagnosis is important not only for treatment and prognostication but also for genetic counselling and antenatal diagnosis in subsequent pregnancies.

DETAILED DESCRIPTION:
Inborn errors of metabolism (IEM) are disorders in which there is a block at some point in the normal metabolic pathway caused by a genetic defect of a specific enzyme. The number of diseases in humans known to be attributable to inherited point defects in metabolism now exceeds 500.While the diseases individually are rare, they collectively account for a significant proportion of neonatal and childhood morbidity and mortality. Diagnosis is important not only for treatment and prognostication but also for genetic counselling and antenatal diagnosis in subsequent pregnancies.So ,the main problems facing the physician caring for a sick newborn infant are to know when to consider the possibility of a metabolic disorder, what to do to determine quickly and efficiently whether a child has a metabolic disease, and how to treat the patient until a diagnosis is established.

One of the clinical presentations that raises red flags of inborn error of metabolism is persistent or recurrent hypoglycemia. However recognizing hypoglycemia in the newborn may be difficult, because the symptoms of hypoglycemia (i.e., lethargy, poor feeding, hypothermia, and seizures) are non specific. Frequent blood sugar determinations are often required to confirm the suspicion of hypoglycemia. Because inborn errors of metabolism are a relatively infrequent cause of neonatal hypoglycemia, other diagnostic possibilities should be investigated concurrently.

The first possibility to consider is neonatal stress secondary to perinatal asphyxia, hypothermia, or intrauterine malnutrition (e.g., placental abnormalities, prematurity, multiple gestations). The second consideration is the possibility of a hormonal abnormality affecting insulin regulation. The inborn errors of metabolism associated with insulin dysregulation include 3-hydroxacyl-CoA dehydrogenase (HADH ) deficiency and hyperammonemia/hyperinsulinism (HA/HI) syndrome, both of which are diazoxide-responsive.The third possibility to consider is a malformation syndrome, specifically including those syndromes associated with hormonal dysregulation such as Beckwith-Wiedemann syndrome. The fourth possibility is that the patient has a severe hepatocellular or cirrhotic liver disease that leads non specifically to fasting hypoglycemia.

Hypoglycemia may be associated with five categories of inborn errors of metabolism: fatty acid oxidation defects gluconeogenesis defects, glycogen storage diseases, ketogenesis defects, and organic acidemias . The diagnostic approach to hypoglycemia, therefore, must give consideration to entities belonging to each of these categories. Usually, Krebs cycle defects and mitochondrial disorders do not produce hypoglycemia, but these defects should be considered when other evidence points in their direction.

The diagnostic approach must quickly narrow the field of possible diagnoses so that specific treatment can be instituted. The classic approaches to the differential diagnosis of hypoglycemic disorders in children are the fasting study and specialized challenge tests. These studies are, however, not feasible in newborn infants because of the significant risks and technical difficulties associated with performing such studies and because of the lack of control data derived from normal neonates. Alternatively, efforts to determine the cause of hypoglycemia in the newborn infant should include hormonal and biochemical studies before and after feeding and especially during an acute episode of hypoglycemia. Definitive diagnosis might have to be postponed several months until the child is old enough to tolerate a formal fasting study or specialized in vitro cell studies.

An algorithm for diagnosing the disorders that cause neonatal hypoglycemia can be generated from the results of the following studies: blood electrolytes and pH, plasma and urinary ketones, plasma free fatty acids, blood lactate and pyruvate, blood ammonia, liver function tests, plasma and urinary carnitine and acylcarnitine analysis, and urinary organic acids. A specific diagnosis might not be made by these studies, but they are necessary for providing a provisional diagnosis that can be confirmed by specific enzyme analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 1day to 28 days .
2. Sex : Both genders .
3. Full Term infant ≥ 37 completed weeks.
4. Persistent hypoglycemia (Blood glucose level ≤ 45 mg/dl/2,5 mmol /L) for more than one reading and not responding to IV fluids and /or oral feeding.

Exclusion Criteria:

1. Age more than 28 days.
2. Newborn with surgical problems.

Ages: 1 Day to 28 Days | Sex: All
Age Groups: Child
Study Population: Any Neonate aged 1 day to 28 days admitted to NICU during one and half year period fulfilling the inclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-10-01 (Estimated); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
Pattern of metabolic diseases in neonates with hypoglycemia | Baseline
  Detection of Pattern of metabolic diseases in neonates with hypoglycemia who admitted to Neonatal Intensive Care Unit NICU at Assiut University Children's Hospital